CLINICAL TRIAL: NCT04039633
Title: Spinal Cord Stimulation for Refractory Pain in Erythromelalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019/159
Record Dates: First submitted 2019-07-30; First posted 2019-07-31 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Erythromelalgia
Keywords: Spinal Cord Stimulation
MeSH Terms: conditions — Erythromelalgia

STUDY DESIGN:
Intervention Model Description: During 6 months following implantation of a pulse generator, all patients will undergo 4 six-week long periods with either burst spinal cord stimulation (SCS) or no stimulation (sham) in a randomized order. During this period all patients will undergo two periods of SCS and sham stimulation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 1st blinding: patients will be blinded to the actual treatment allocation during the different study periods (first blinding). 2nd: surgeons and all study personnel involved in handling the patients and collecting the study data (except those who perform the actual setting of the device) will be blinded to the actual treatment allocation. 3rd: All study personnel evaluating end point measures will be blinded to the actual treatment. 4th All the tables and figures to be presented from the study will be settled before any data from the study is evaluated in order to avoid selective presentation of findings according to statistical results. 5th The statistician performing the statistical procedures on the outcome of the study will be blinded. The data will only show treatment allocation as treatment A and treatment B. Then the tables and figures are filled in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Burst spinal cord stimulation (SCS) (Experimental): following implantation of a generator that sends pulses to a thin wire (lead), which delivers pulses to nerves along the spinal cord, the patients will initially undergo four six-week long periods with either burst SCS or no stimulation (sham) in a randomized order. During this period all patients will undergo two periods of SCS and sham stimulation.
  Interventions: Procedure: Burst Spinal Cord Stimulation; Procedure: Sham spinal cord stimulation
- sham spinal cord stimulation (SCS) (Sham Comparator): following implantation of a generator that sends pulses to a thin wire (lead), which delivers pulses to nerves along the spinal cord, the patients will initially undergo four six-week long periods with either burst SCS or no stimulation (sham) in a randomized order. During this period all patients will undergo two periods of SCS and sham stimulation.
  Interventions: Procedure: Burst Spinal Cord Stimulation; Procedure: Sham spinal cord stimulation

INTERVENTIONS:
Procedure: Burst Spinal Cord Stimulation — Burst stimulation utilizes complex programming to deliver high-frequency stimuli of a 40 Hz burst mode with 5 spikes at 500 Hz per spike delivered in a constant current mode
Procedure: Sham spinal cord stimulation — A pulse generator is implanted, but no spinal cord stimulation is provided

SUMMARY:
Erythromelalgia is a rare disorder characterized by red, warm, and painful extremities, which is often precipitated by warm conditions. The pathophysiology is incompletely understood. The management of pain in erythromelalgia is challenging as no single therapy has been found to be effective. Response to pharmacotherapy varies, meaning that the physician has to take a stepwise trial and error approach with each patient. Consequently, this disorder is often associated with poorer health-related quality of life. There is currently no consensus or guideline on management of pain in erythromelalgia. Spinal cord stimulation is a widely applied therapy to treat severe chronic pain of various origin. Case reports and anecdotal evidence suggest that this therapy might alleviate refractory pain in patients with erythromelalgia.

The aim of this trial is to evaluate the efficacy of spinal cord stimulation for refractory pain in erythromelalgia.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of primary or idiopathic erythromelalgia
2. Patients ≥18 years who have developed chronic pain that has remained refractory to medical treatment for ≥6 months.
3. Minimum pain intensity of 5/10 on a numeric rating scale NRS at baseline.
4. Successful two-week SCS testing period with tonic stimulation (≥2 points reduction in pain NRS from baseline). This means patients will experience paresthesia during the trial period of spinal cord stimulation.

Exclusion Criteria:

1. Coexisting conditions that would increase procedural risk (e.g., sepsis, coagulopathy).
2. History of laminectomy or posterior fusion at the thoracolumbar junction, where percutaneous electrode end tips are routinely placed.
3. Abnormal pain behavior and/or unresolved psychiatric illness.
4. Unresolved issues of secondary gain or inappropriate medication use.
5. Unfit for participation for any other reason as judged by the study physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Changes in pain | 6 months
  assessed with a 0 -to-10 numerical rating scale (NRS)

SECONDARY OUTCOMES:
Change in generic health-related quality of life | 6 months
  Assessed with the Euro-Qol-5D (5L)
Oswestry disability index (ODI) score | 6 months
  questionnaire originally designed to quantify disability for degenerative conditions of the lumbar spine, possibly a relevant outcome measure also in patients with erythromelalgia as it covers intensity of pain, ability to care for oneself, ability to walk, ability to sit, ability to lift, sexual function, ability to stand, social life, sleep quality, and ability to travel. The index is scored from 0 to 100. Zero means no disability and 100 reflects maximum disability.
Daily physical activity | 6 months
  measured by use of a body-worn accelerometer (activPALs from PAL Technologies Ltd., Glasgow, United Kingdom) attached by a waterproof tape to the midpoint of the patients' anterior right thigh
Severity of erythema | 6 months
  assessed using the Patient's Self-Assessment (PSA) scale
Health Care Provider's Costs | 6 months
  Cost-effectiveness (cost per gained quality-adjusted life year)

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Gulati, md prof, Principal Investigator — St. Olavs Hospital; Geir Bråthen, md prof, Study Director — St. Olavs Hospital
Locations (4):
- Norway (4):
  - Halden Dermatology Center, Halden
  - Aleris, Strømmen
  - Universitetssykehuset nord-norge hf, Tromsø
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473